CLINICAL TRIAL: NCT02097121
Title: BOTOX® in the Treatment of Urinary Incontinence Due to Overactive Bladder in Patients 12 to 17 Years of Age
Brief Title: OnabotulinumtoxinA for the Treatment of Urinary Incontinence Due to Overactive Bladder in Pediatric Patients (12 to 17)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-137; 2014-000464-17 (EudraCT Number)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Urinary Incontinence; Urinary Bladder; Overactive
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Botox 25 U (Experimental): Participants randomized to receive 25 Units (U) BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone. Posttreatment follow-up clinic visits occurred at Weeks 2, 6, and 12. Participants could request retreatment from Week 12 and 12 weeks after each subsequent treatment for up to 4 cycles. The retreatment dose was determined by the Investigator and could be at the same dose or at the next higher dose compared with the preceding treatment.
  Interventions: Biological: BOTOX®
- Botox 50 U (Experimental): Participants randomized to receive 50 Units (U) BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone. Posttreatment follow-up clinic visits occurred at Weeks 2, 6, and 12. Participants could request retreatment from Week 12 and 12 weeks after each subsequent treatment for up to 4 cycles. The retreatment dose was determined by the Investigator and could be at the same dose or at the next higher dose compared with the preceding treatment.
  Interventions: Biological: BOTOX®
- Botox 100 U (Experimental): Participants randomized to receive 100 Units (U) BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone. Posttreatment follow-up clinic visits occurred at Weeks 2, 6, and 12. Participants could request retreatment from Week 12 and 12 weeks after each subsequent treatment for up to 4 cycles. The retreatment dose was determined by the Investigator and could be at the same dose or at the next higher dose compared with the preceding treatment.
  Interventions: Biological: BOTOX®

INTERVENTIONS:
Biological: BOTOX® — Each vial of BOTOX (Botulinum Toxin Type A) purified neurotoxin complex, formulation No. 9060X contains 100 U of Clostridium botulinum toxin Type A, 0.5 mg albumin (human), and 0.9 mg sodium chloride in a sterile, vacuum-dried form without a preservative. The study medication was to be reconstituted with 0.9% sodium chloride (preservative-free). The 10 mL of study drug was to be administered as 20 injections each of 0.5 mL. Under direct cystoscopic visualization, injections were to be distributed evenly across the detrusor wall and spaced approximately 1 cm apart. To avoid injecting the trigone, the injections were to be at least 1 cm above the trigone. The injection needle was to be inserted approximately 2 mm into the detrusor for each injection.
  Other Names: Botulinum Toxin Type A

SUMMARY:
This was a multicenter, randomized, double-blind, parallel-group, multiple-dose study to evaluate the efficacy and safety of BOTOX in adolescents with urinary incontinence due to overactive bladder (OAB) with inadequate management with anticholinergic therapy. Participants were randomized in a 1:1:1 ratio to receive a single Tx of 25 U, 50 U, or 100 U BOTOX (not to exceed 6 U/kg) on Day 1, were seen after each treatment at Weeks 2, 6, and 12 post-treatment, and thereafter at alternating telephone and clinic visits every 6 weeks until they qualified for further retreatment/exited the study. Participants could receive multiple treatments dependent upon the number and timing of patient requests/qualification for retreatment. At each retreatment the investigator could keep the dose the same or increase it one dose level in a blinded fashion. Participants exited the study once 96 weeks have elapsed since entry on Day 1 and at least 12 weeks follow-up since their last study treatment had occurred.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder (OAB) (frequency/urgency) with urinary incontinence for at least 6 months
* OAB symptoms not adequately managed by 1 or more anticholinergic agents

Exclusion Criteria

* OAB caused by a neurological condition
* Use of anticholinergics or other medications to treat OAB symptoms within 7 days
* Current use of indwelling catheter or clean intermittent catheterization to empty the bladder
* Previous or current use of botulinum toxin therapy of any serotype for any urological condition, or treatment with botulinum toxin of any serotype within 3 months for any other condition or use
* Myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (39):
- United States (8):
  - Alaska Urological Institute /ID# 238189, Anchorage, Alaska
  - Arkansas Children's Hospital /ID# 237787, Little Rock, Arkansas
  - Children's Hospital Colorado /ID# 237621, Aurora, Colorado
  - Yale New Haven Hospital - Yale School of Medicine /ID# 238222, New Haven, Connecticut
  - Orlando Health-Arnold Palmer Hospital for Children Pediatric Urology /ID# 235283, Orlando, Florida
  - Associated Urologist of North Carolina /ID# 235437, Raleigh, North Carolina
  - Cook Children's Med. Center /ID# 237539, Fort Worth, Texas
  - Children's Hospital Wisconsin - Milwaukee Campus /ID# 237544, Milwaukee, Wisconsin
- Australia (3):
  - Sydney Children's Hospital /ID# 237191, Randwick, New South Wales
  - The Children's Hospital at Westmead /ID# 234337, Sydney, New South Wales
  - Monash Children's Hospital /ID# 234388, Clayton, Victoria
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen /ID# 237997, Edegem, Antwerpen
  - UZ Gent /ID# 237588, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 237218, Leuven, Vlaams-Brabant
- Canada (3):
  - Alberta Children's Hospital /ID# 237510, Calgary, Alberta
  - London Health Sciences Center /ID# 234304, London, Ontario
  - CHUS - Hopital Fleurimont /ID# 237668, Sherbrooke, Quebec
- Fakultni nemocnice Olomouc /ID# 237577, Olomouc, Czechia
- France (3):
  - Duplicate_CHU Bordeaux-Hopital Pellegrin /ID# 237392, Bordeaux
  - Hôpital de la Mère et de l'Enfant /ID# 235227, Limoges
  - Hôpitaux Pédiatriques de Nice CHU-LENVAL /ID# 235278, Nice
- Germany (3):
  - Evangelisches Krankenhaus Bielefeld /ID# 235234, Bielefeld
  - Urologische Gemeinschaftspraxis /ID# 234978, Emmendingen
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 234288, Lübeck
- AOU Universita degli Studi della Campania Luigi Vanvitelli /ID# 237308, Napoli, Italy
- Netherlands (2):
  - Radboud Universitair Medisch Centrum /ID# 237043, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum /ID# 237678, Maastricht
- Oslo University Hospital /ID# 234434, Oslo, Norway
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu /ID# 238166, Wroclaw, Lower Silesian Voivodeship
  - Specjalistyczny Gabinet Lekarski /ID# 235257, Poznan
  - Medical Concierge Centrum Medyczne /ID# 235200, Warsaw
- St Georges Hospital /ID# 235316, Port Elizabeth, South Africa
- United Kingdom (7):
  - Manchester University NHS Foundation Trust /ID# 234380, Manchester, Lancashire
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 234819, Norwich, Norfolk
  - NHS Greater Glasgow and Clyde /ID# 237430, Glasgow, Scotland
  - NHS Grampian /ID# 237379, Aberdeen
  - Alder Hey Children's NHS Foundation Trust /ID# 237279, Liverpool
  - Royal Berkshire NHS Foundation Trust /ID# 236915, Reading
  - Sheffield Children's NHS Foundation Trust /ID# 237854, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com.,To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to 1 of 3 treatment arms. Randomization was stratified by baseline daytime urinary urgency incontinence episodes (a total of ≤ 6 episodes or > 6 episodes over the 2-day bladder diary collection period).
Period: Overall Study
Arm/Group | Botox 25 U | Botox 50 U | Botox 100 U
Started | 19 | 18 | 19
Received Any Treatment | 19 | 17 | 19
Actual Treatment Received in Cycle 1 | 18 | 17 | 20 (One participant randomized to 25 U BOTOX received 100 U BOTOX in Cycle 1 in error)
Actual Treatment Received in Cycle 2 | 1 | 17 (One participant assigned to 100 U BOTOX received 50 U BOTOX in Cycle 2 in error) | 28 (One participant assigned to 25 U BOTOX and two participants assigned to 50 U BOTOX received 100 U BOTOX in Cycle 2 in error)
Actual Treatment Received in Cycle 3 | 2 | 7 | 13
Actual Treatment Received in Cycle 4 | 0 | 1 | 3
Completed | 12 | 12 | 9
Not Completed | 7 | 6 | 10
Not completed — Other, not specified | 4 | 2 | 3
Not completed — Lack of Efficacy | 2 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The BOTOX-treated population (all participants enrolled into the study who received at least 1 BOTOX treatment) according to the dose received in the first treatment cycle.
Groups:
- BOTOX 25 U (BOTOX-Treated Population): Participants received 25 U BOTOX in Treatment Cycle 1
- BOTOX 50 U (BOTOX-Treated Population): Participants received 50 U BOTOX in Treatment Cycle 1
- BOTOX 100 U (BOTOX-Treated Population): Participants received 100 U BOTOX in Treatment Cycle 1
- Total: Total of all reporting groups
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population) | Total
Number analyzed (Participants) | 18 | 17 | 20 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 17 | 20 | 55
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.49) | 14.3 (1.86) | 14.0 (1.75) | 14.0 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 14 | 47
  Male | 2 | 0 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 17 | 41
  Black or African American | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Hispanic | 0 | 0 | 0 | 0
  Other | 1 | 1 | 1 | 3
  Not reported | 2 | 1 | 1 | 4
  Unknown | 3 | 2 | 1 | 6
Daily Frequency of Daytime Urinary Incontinence Episodes [Mean (Standard Deviation); unit: number of episodes] — A bladder diary was used to log each daytime urgency episode over 2 consecutive days during screening.
  number of episodes | 5.29 (3.447) | 3.54 (2.696) | 3.64 (2.951) | 4.15 (3.100)

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in the Daily Normalized Daytime Average Number of Urinary Incontinence Episodes in Treatment Cycle 1
Description: Urinary incontinence was defined as involuntary loss of urine as recorded by the participant in a bladder diary during 2 consecutive days in the week prior to the study visit (normalized to a 12 hour daytime period). Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. The number of daily daytime incontinence episodes were averaged during the 2-day period. A negative change from Baseline indicates improvement. Data are summarized per the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: From Baseline to 2 consecutive days in the week prior to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: urinary incontinence episodes per day
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
urinary incontinence episodes per day | -1.37 (0.801) | -0.97 (0.811) | -2.35 (0.746)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); Treatment Difference of 100 U versus 25 U Pairwise comparisons of 100 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using an ANCOVA model with study baseline value as covariate, and treatment group as factor. A hierarchical analysis strategy to adjust for multiplicity was used; Test type: Superiority; p = 0.3802, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-3.203 to 1.243], Standard Error of Mean 1.107
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); Treatment Difference of 50 U versus 25 U Pairwise comparisons of 50 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using an ANCOVA model with study baseline value as covariate, and treatment group as factor. A hierarchical analysis strategy to adjust for multiplicity was used; Test type: Superiority; p = 0.733, ANCOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-1.921 to 2.712], Standard Error of Mean 1.154

2. Secondary Outcome: Change From Study Baseline in the Daily Average Frequency of Normalized Daytime Micturition Episodes
Description: Micturition was defined as toilet voids recorded by the participant in a bladder diary during 2 consecutive days in the week prior to the study visit (normalized to a 12 hour daytime period). Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. The number of daily daytime micturition episodes were averaged during the 2-day period. A negative change from Baseline indicates improvement. Data are summarized per the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: From Baseline to 2 consecutive days in the week prior to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: micturition episodes per day
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
micturition episodes per day | -1.84 (1.027) | 0.31 (1.014) | -1.02 (0.983)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); Treatment Difference of 100 U versus 25 U Pairwise comparisons of 100 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using an ANCOVA model with study baseline value as covariate, and treatment group and stratification (baseline daytime urinary urgency incontinence episodes [a total of ≤ 6 episodes or > 6 episodes over the 2-day diary collection period]) as factors. A hierarchical analysis strategy to adjust for multiplicity was not implemented; Test type: Superiority; p = 0.5743, ANCOVA; LS Mean Difference = 0.82, 95% CI 2-sided [-2.082 to 3.713], Standard Error of Mean 1.442
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); Treatment Difference of 50 U versus 25 U Pairwise comparisons of 50 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using an ANCOVA model with study baseline value as covariate, and treatment group and stratification (baseline daytime urinary urgency incontinence episodes [a total of ≤ 6 episodes or > 6 episodes over the 2-day diary collection period]) as factors. A hierarchical analysis strategy to adjust for multiplicity was not implemented; Test type: Superiority; p = 0.1451, ANCOVA; LS Mean Difference = 2.15, 95% CI 2-sided [-0.769 to 5.078], Standard Error of Mean 1.455

3. Secondary Outcome: Change From Study Baseline in the Daily Average Frequency of Normalized Daytime Urgency Episodes
Description: Participants recorded daytime urgency episodes in a bladder diary during 2 consecutive days in the week prior to the study visit (normalized to a 12 hour daytime period). Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. The number of daily daytime urgency episodes were averaged during the 2-day period. A negative change from Baseline indicates improvement. Data are summarized per the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: From Baseline to 2 consecutive days in the week prior to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: urgency episodes per day
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
urgency episodes per day | -1.85 (1.014) | -1.78 (0.998) | -2.18 (0.945)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8206, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-3.205 to 2.551], Standard Error of Mean 1.434
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.9604, ANCOVA; LS Mean Difference = 0.07, 95% CI 2-sided [-2.807 to 2.95], Standard Error of Mean 1.434

4. Secondary Outcome: Percentage of Participants With Night Time Urinary Incontinence
Description: Urinary incontinence was defined as involuntary loss of urine. Participants recorded night time urinary incontinence episodes in a bladder diary during 2 consecutive days in the week prior to the study visit. Night time is defined as the time between going to bed to sleep for the night and waking up to start the next day. The number of daily night time urinary incontinence episodes were averaged during the 2-day period. Data are summarized per the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: From Baseline to 2 consecutive days in the week prior to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
percentage of participants
  Baseline-0 nights | 22.2 | 52.9 | 35.0
  Baseline-1 night | 27.8 | 11.8 | 15.0
  Baseline-2 nights | 50.0 | 35.3 | 50.0
  Week 12-0 nights | 50.0 | 76.5 | 50.0
  Week 12-1 night | 22.2 | 5.9 | 15.0
  Week 12-2 nights | 27.8 | 17.6 | 35.0

5. Secondary Outcome: Change From Study Baseline in the Daily Average Volume Voided Per Micturition (mL)
Description: The volume per micturition was derived from the total urine volume voided over 1 daytime period during the 2-day bladder diary collection period divided by the number of voids in the same daytime period. Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. A negative change from Baseline indicates improvement. Data are summarized per the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: From Baseline to 2 consecutive days in the week prior to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
mL | -9.17 (15.924) | 24.94 (17.047) | 26.16 (15.900)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1174, ANCOVA; LS Mean Difference = 35.33, 95% CI 2-sided [-9.207 to 79.873], Standard Error of Mean 22.175
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.1567, ANCOVA; LS Mean Difference = 34.11, 95% CI 2-sided [-13.536 to 81.76], Standard Error of Mean 23.722

6. Secondary Outcome: Change From Study Baseline in Pediatric Urinary Incontinence Quality of Life Total Score (PinQ)
Description: The PinQ is a 20-item questionnaire that asks about the participant's incontinence and its consequences in daily life and relationships. Items are answered on a Likert-type scale of 0 (no) to 4 (all of the time) and a total sum score is calculated (from 0 to 80), with higher scores indicating lower health-related quality of life. A negative change from Baseline indicates improvement.
Time Frame: From Day 1 Prior to Treatment to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
units on a scale | -6.96 (2.841) | -5.11 (3.243) | -8.28 (2.979)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7481, ANCOVA; LS Mean Difference = -1.32, 95% CI 2-sided [-9.553 to 6.909], Standard Error of Mean 4.091
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.6691, ANCOVA; LS Mean Difference = 1.85, 95% CI 2-sided [-6.799 to 10.498], Standard Error of Mean 4.299

7. Secondary Outcome: Change From Study Baseline in PinQ Item 'I am Worried That People Might Think my Clothes Smell Like Pee"
Description: The Pediatric Urinary Incontinence Quality of (PinQ) is a 20-item questionnaire that asks about the participant's incontinence and its consequences in daily life and relationships. Items are answered on a Likert-type scale of 0 (no) to 4 (all of the time), with higher scores indicating lower health-related quality of life. A negative change from Baseline indicates improvement.
Time Frame: From Day 1 Prior to Treatment to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
units on a scale | -0.06 (0.238) | -0.37 (0.273) | -0.09 (0.251)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9297, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.721 to 0.661], Standard Error of Mean 0.343
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); Pairwise comparisons of 50 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using an ANCOVA model with study baseline value as covariate, and treatment group and stratification (baseline daytime urinary urgency incontinence episodes [a total of ≤ 6 episodes or > 6 episodes over the 2-day diary collection period]) as factors. A hierarchical analysis strategy to adjust for multiplicity was not implemented; Test type: Superiority; p = 0.3976, ANCOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-1.022 to 0.413], Standard Error of Mean 0.357

8. Secondary Outcome: Change From Study Baseline in PinQ Item 'My Bladder Problem Makes me Feel Bad About Myself"
Description: as for outcome 7
Time Frame: From Day 1 Prior to Treatment to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
units on a scale | -0.54 (0.209) | -0.15 (0.238) | -0.24 (0.220)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3309, ANCOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.311 to 0.904], Standard Error of Mean 0.302
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.2235, ANCOVA; LS Mean Difference = 0.39, 95% CI 2-sided [-0.245 to 1.024], Standard Error of Mean 0.315

9. Secondary Outcome: Change From Study Baseline in PinQ Item 'I Miss Out on Being With Friends Because of my Bladder Problems"
Description: as for outcome 7
Time Frame: From Day 1 Prior to Treatment to Week 12 in Treatment Cycle 1
Population: Participants with analysis values at both baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 20
units on a scale | -0.39 (0.193) | -0.24 (0.218) | -0.27 (0.201)
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6689, ANCOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-0.434 to 0.67], Standard Error of Mean 0.274
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.6076, ANCOVA; LS Mean Difference = 0.15, 95% CI 2-sided [-0.431 to 0.729], Standard Error of Mean 0.288

10. Secondary Outcome: Percentage of Participants With a Positive Treatment Response in the Modified Treatment Benefit Scale
Description: The Modified Treatment Benefit Scale (Modified TBS) is a single-item scale designed to assess the change in the participant's overactive bladder (OAB) condition following treatment. The participant's current condition (urinary problems, urinary incontinence) is compared to their condition prior to receipt of any study treatment by selection of "greatly improved", "improved", "not changed" or "worsened". Participants who selected "greatly improved" or "improved" were considered to have a positive treatment response.
Time Frame: At Week 12 in Treatment Cycle 1
Population: Participants with non-missing values at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 17 | 17 | 19
percentage of participants | 52.9 [27.81 to 77.02] | 70.6 [44.04 to 89.69] | 68.4 [43.45 to 87.42]
Statistical Analysis 1: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 100 U (BOTOX-Treated Population); Treatment Difference of 100 U versus 25 U Pairwise comparisons of 100 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using the Cochran-Mantel-Haenszel (CMH) method stratified by baseline daytime urinary urgency incontinence episodes (a total of ≤ 6 episodes or > 6 episodes over the 2-day diary collection period); Test type: Superiority; p = 0.6092, Cochran-Mantel-Haenszel; Risk difference % = 15.5, 95% CI 2-sided [-18.94 to 46.19]
Statistical Analysis 2: Comparison: BOTOX 25 U (BOTOX-Treated Population) vs BOTOX 50 U (BOTOX-Treated Population); Treatment Difference of 50 U versus 25 U Pairwise comparisons of 50 U versus 25 U of BOTOX up to Week 12 in Treatment Cycle 1 was evaluated using the Cochran-Mantel-Haenszel (CMH) method stratified by baseline daytime urinary urgency incontinence episodes (a total of ≤ 6 episodes or > 6 episodes over the 2-day diary collection period); Test type: Superiority; p = 0.4824, Cochran-Mantel-Haenszel; Risk difference % = 17.6, 95% CI 2-sided [-16.2 to 48.9]

11. Secondary Outcome: Time to Participant's First Request for Retreatment
Description: The time from the day of BOTOX treatment to the request for the subsequent treatment was estimated using a Kaplan-Meier survival method for each treatment group. Participants who did not request retreatment were treated as censored at the time of their last study visit or study exit.
Time Frame: From the day of BOTOX treatment in Treatment Cycle 1 to the request for subsequent treatment
Population: BOTOX-treated participants who requested retreatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 17 | 14 | 17
weeks | 16.6 [12.71 to 25.29] | 17.6 [11.29 to 38.57] | 21.3 [12.86 to 30.14]

12. Secondary Outcome: Time to Participant's Qualification for Retreatment
Description: The time from the day of BOTOX treatment to the qualification for retreatment was estimated using a Kaplan-Meier survival method for each treatment group. Participants who did not qualify for retreatment were treated as censored at the time of their last study visit or study exit.
Time Frame: From the day of BOTOX treatment in Treatment Cycle 1 to the qualification for retreatment
Population: BOTOX-treated participants who qualified for retreatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 16 | 14 | 17
weeks | 22.5 [13.57 to 36.29] | 18.1 [12.29 to 52.57] | 24.1 [12.86 to 41.57]

13. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From the first dose of study drug until the last dose, up to 147 weeks
Population: All participants enrolled into the study who received at least 1 BOTOX treatment
Measure: Count of Participants; unit: Participants
Groups:
- BOTOX 25 U (BOTOX-Treated Population): Participants received 25 U BOTOX in a given Treatment Cycle
- BOTOX 50 U (BOTOX-Treated Population): Participants received 50 U BOTOX in a given Treatment Cycle
- BOTOX 100 U (BOTOX-Treated Population): Participants received 100 U BOTOX in a given Treatment Cycle
Arm/Group | BOTOX 25 U (BOTOX-Treated Population) | BOTOX 50 U (BOTOX-Treated Population) | BOTOX 100 U (BOTOX-Treated Population)
Number analyzed (Participants) | 18 | 17 | 28
Participants
  Cycle 1: number analyzed (Participants) | 18 | 17 | 20
  Cycle 1 | 13 | 12 | 14
  Cycle 2: number analyzed (Participants) | 1 | 17 | 28
  Cycle 2 | 1 | 13 | 18
  Cycle 3: number analyzed (Participants) | 2 | 7 | 13
  Cycle 3 | 1 | 3 | 8
  Cycle 4: number analyzed (Participants) | 0 | 1 | 3
  Cycle 4 |  | 1 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study; median time on follow-up was up to 724 days. TEAEs/SAEs were collected from the first dose of study drug until the last dose, up to 147 weeks.
Description: For safety analyses, participants were assigned to a treatment group based on the treatment actually received, regardless of the treatment randomized.
Groups:
- 25 U BOTOX All: All participants who received 25 U BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 50 U BOTOX All: All participants who received 50 U BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 100 U BOTOX All: All participants who received 100 U BOTOX (not to exceed 6 U/kg), administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 25 U BOTOX Cycle 1: Participants who received 25 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 1, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 50 U BOTOX Cycle 1: Participants who received 50 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 1, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 100 U BOTOX Cycle 1: Participants who received 100 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 1, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- All BOTOX Cycle 1: All BOTOX-treated participants in Treatment Cycle 1
- 25 U BOTOX Cycle 2: Participants who received 25 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 2, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 50 U BOTOX Cycle 2: Participants who received 50 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 2, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 100 U BOTOX Cycle 2: Participants who received 100 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 2, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- All BOTOX Cycle 2: All BOTOX-treated participants in Treatment Cycle 2
- 25 U BOTOX Cycle 3: Participants who received 25 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 3, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 50 U BOTOX Cycle 3: Participants who received 50 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 3, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 100 U BOTOX Cycle 3: Participants who received 100 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 3, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- All BOTOX Cycle 3: All BOTOX-treated participants in Treatment Cycle 3
- 25 U BOTOX Cycle 4: Participants who received 25 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 4, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 50 U BOTOX Cycle 4: Participants who received 50 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 4, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- 100 U BOTOX Cycle 4: Participants who received 100 U BOTOX (not to exceed 6 U/kg) in Treatment Cycle 4, administered via cystoscopy as 20 intradetrusor injections of 0.5 mL each, sparing the trigone.
- All BOTOX Cycle 4: All BOTOX-treated participants in Treatment Cycle 4
Arm/Group | 25 U BOTOX All | 50 U BOTOX All | 100 U BOTOX All | 25 U BOTOX Cycle 1 | 50 U BOTOX Cycle 1 | 100 U BOTOX Cycle 1 | All BOTOX Cycle 1 | 25 U BOTOX Cycle 2 | 50 U BOTOX Cycle 2 | 100 U BOTOX Cycle 2 | All BOTOX Cycle 2 | 25 U BOTOX Cycle 3 | 50 U BOTOX Cycle 3 | 100 U BOTOX Cycle 3 | All BOTOX Cycle 3 | 25 U BOTOX Cycle 4 | 50 U BOTOX Cycle 4 | 100 U BOTOX Cycle 4 | All BOTOX Cycle 4
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/29 | 0/33 | 0/18 | 0/17 | 0/20 | 0/55 | 0/1 | 0/17 | 0/28 | 0/46 | 0/2 | 0/7 | 0/13 | 0/22 | 0/0 | 0/1 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/29 | 1/33 | 1/18 | 0/17 | 0/20 | 1/55 | 0/1 | 0/17 | 1/28 | 1/46 | 0/2 | 0/7 | 1/13 | 1/22 | 0/0 | 0/1 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 12/18 | 23/29 | 24/33 | 12/18 | 12/17 | 14/20 | 38/55 | 1/1 | 13/17 | 18/28 | 32/46 | 1/2 | 3/7 | 8/13 | 12/22 | 0/0 | 1/1 | 1/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 U BOTOX All (N=18) | 50 U BOTOX All (N=29) | 100 U BOTOX All (N=33) | 25 U BOTOX Cycle 1 (N=18) | 50 U BOTOX Cycle 1 (N=17) | 100 U BOTOX Cycle 1 (N=20) | All BOTOX Cycle 1 (N=55) | 25 U BOTOX Cycle 2 (N=1) | 50 U BOTOX Cycle 2 (N=17) | 100 U BOTOX Cycle 2 (N=28) | All BOTOX Cycle 2 (N=46) | 25 U BOTOX Cycle 3 (N=2) | 50 U BOTOX Cycle 3 (N=7) | 100 U BOTOX Cycle 3 (N=13) | All BOTOX Cycle 3 (N=22) | 25 U BOTOX Cycle 4 (N=0) | 50 U BOTOX Cycle 4 (N=1) | 100 U BOTOX Cycle 4 (N=3) | All BOTOX Cycle 4 (N=4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOCIAL PROBLEM (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALLOR (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 U BOTOX All (N=18) | 50 U BOTOX All (N=29) | 100 U BOTOX All (N=33) | 25 U BOTOX Cycle 1 (N=18) | 50 U BOTOX Cycle 1 (N=17) | 100 U BOTOX Cycle 1 (N=20) | All BOTOX Cycle 1 (N=55) | 25 U BOTOX Cycle 2 (N=1) | 50 U BOTOX Cycle 2 (N=17) | 100 U BOTOX Cycle 2 (N=28) | All BOTOX Cycle 2 (N=46) | 25 U BOTOX Cycle 3 (N=2) | 50 U BOTOX Cycle 3 (N=7) | 100 U BOTOX Cycle 3 (N=13) | All BOTOX Cycle 3 (N=22) | 25 U BOTOX Cycle 4 (N=0) | 50 U BOTOX Cycle 4 (N=1) | 100 U BOTOX Cycle 4 (N=3) | All BOTOX Cycle 4 (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MISOPHONIA (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC FATIGUE SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILLNESS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIURIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (4) | 6 (8) | 1 (1) | 2 (4) | 3 (4) | 6 (9) | 0 (0) | 0 (0) | 4 (6) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 6 (11) | 6 (9) | 2 (3) | 2 (4) | 2 (5) | 6 (12) | 0 (0) | 4 (7) | 9 (12) | 13 (19) | 0 (0) | 2 (3) | 4 (5) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL DISCOMFORT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CRYSTAL URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPSTEIN-BARR VIRUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESIDUAL URINE VOLUME (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URINE LEUKOCYTE ESTERASE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ABNORMAL WEIGHT GAIN (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SACRAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANOREXIA NERVOSA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER DISCOMFORT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 2 (2) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 4 (4) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOCYTURIA (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETHRAL PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA GENITAL (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (2) | 1 (1) | 1 (3) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL BED INFLAMMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2014-09-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02097121/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02097121/SAP_001.pdf